CLINICAL TRIAL: NCT02008084
Title: A Randomized, Double-blind, Placebo-controlled, Forced Dose-escalation, Multi-center Pilot Study to Evaluate the Lipid Regulating Effects of TRIA-662 (1-methylnicotinamide Chloride)
Brief Title: A Pilot Study to Evaluate the Lipid Effects of TRIA-662
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cortria Corporation (Industry)
Collaborators: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PNAI-MNA-03
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Hypertriglyceridemia; Mixed Hyperlipidemia
Keywords: hypertriglyceridemia; mixed hyperlipidemia
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TRIA-662 single-blind baseline (Sham Comparator): Baseline, 6 to 8-week, dietary lead-in period
  Interventions: Drug: TRIA-662; Drug: Placebo
- TRIA-662 (Experimental): Following successful completion of the Baseline randomized to active drug
  Interventions: Drug: TRIA-662
- Placebo (Placebo Comparator): Following successful completion of the Baseline randomized to placebo drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRIA-662 — Following Baseline randomized to active TRIA-662 2 x 500 mg tablets, three times daily with meals for 2 weeks and then active TRIA-662 2 x 1000 mg tablets, three times daily with meals for 12 weeks.
  Arms: TRIA-662; TRIA-662 single-blind baseline
Drug: Placebo — Following Baseline randomized to placebo TRIA-662 2 x 500 mg tablets, three times daily with meals for 2 weeks and then placebo TRIA-662 2 x 1000 mg tablets, three times daily with meals for 12 weeks.
  Arms: Placebo; TRIA-662 single-blind baseline

SUMMARY:
The purpose of this pilot study is to learn what study factors are important in designing a large, full-scale study of the effects of TRIA-662 on serum triglycerides (TG) and high-density lipoprotein cholesterol (HDL-C) levels. In this study, patients will first enter a Single-blind, dietary-controlled baseline period and receive 1000 mg placebo or active drug three times daily with meals (i.e., breakfast, lunch, and dinner) for 6 - 8 weeks. If the qualify to continue, they will then receive up to 2000 mg of active or placebo drug for an additional 14 weeks. Active drug will be given to 48 patients and placebo drug will be given to 16 patients. However, neither the patients not the clinic staff will know which patients are on active or placebo drug until the end of the study.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess the feasibility of a large,full-scale study that would evaluate the regulating effects of TRIA-662 on serum triglycerides (TG) and high-density lipoprotein cholesterol (HDL-C) levels. In this study, patients will first enter a Single-blind, dietary-controlled baseline period and receive 1000 mg placebo or active drug three times daily with meals (i.e., breakfast, lunch, and dinner) for 6 - 8 weeks. Upon completion of the 6 to 8 -week dietary-controlled baseline period, subjects meeting all inclusion and no exclusion criteria will be randomized to the double-blind treatment period. In the double-blind treatment period patients will be randomized such that at least 48 subjects will be randomized to TRIA-662 and at least 16 patients will be randomized to placebo (3:1 ratio). The forced-dose titration will be achieved as follows: Weeks 1 - 2: Two 500 mg tablets three times daily with meals (total daily dose 3000 mg); Weeks 3 - 14: Two 1000 mg tablets three times daily with meals (total daily dose 6000 mg).

Investigational product will be administered three times daily with meals (i.e., breakfast, lunch, and dinner). Down titration to 3000 mg daily (two 500 mg tablets, three times daily) is allowed in the event that a patient cannot tolerate the 6000 mg daily treatment for the stipulated period. Under this scenario, the down-titrated patient will remain on the tolerated dose for the remainder of the study. Lipid and ancillary exploratory parameters will be evaluated during the baseline period, upon randomization and throughout the active treatment period. Throughout the study, patients must adhere to a heart-healthy diet, abstain from/minimize ethyl alcohol intake and control any other variables that may alter serum lipid levels (e.g., exercise, weight loss programs, drugs including over the counter agents preparations that may alter serum lipid levels. Safety and tolerability will be assessed throughout the trial through the evaluation of physical exams, electrocardiograms (ECGs), routine hematology and blood chemistry testing, vital signs and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Women of childbearing potential must have a negative serum pregnancy test at screening and Visit 4

   Women are considered not of childbearing potential if they:
   1. have had a hysterectomy or tubal ligation prior to Visit 1.
   2. are postmenopausal (12 months no menses or menopausal follicle stimulating hormone level) Women of childbearing potential must agree to use an effective method of birth control throughout the study. Acceptable means of birth control include: implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, male or female condoms with spermicide, abstinence, or a sterile sexual partner.
2. Patients who at Weeks -4 and -2 demonstrate mean LDL-C at the levels at which lipid-modifying drug therapy is not indicated according to investigator judgment under ATP III guidelines.
3. Patients who demonstrate mean serum triglycerides = or >200 mg/dL (2.26 mmol/L) but < or = 500 mg/dL (5.65 mmol/L) as measured at 2 sequential visits during the dietary controlled baseline period (Visits 2 and 3 or Visits 3 and 3a) and having lower level within 25% of upper level (higher value minus lower value)/higher value < 0.25).
4. Patients willing to maintain a stable diet and physical activity level throughout the study
5. Patients willing and able to sign the information and consent form and follow the protocol including availability for all visits/telephone follow-up for approximately 24 weeks.

Exclusion Criteria:

1. pregnant, planning to become pregnancy during the study, or nursing
2. clinically significant electrocardiographic abnormalities at Visit 1 or 4
3. body mass index > 45 kg/m2 at Visit 1
4. weight change of > 5% of initial body weight between Visit 1 and 4
5. poorly controlled diabetes defined as a hemoglobin A1c > 9.5% prior to Visit 4
6. evidence of hepatic disease (ALT or AST greater than 2.0 upper limit of normal (ULN), bilirubin > 1.5 ULN, or cirrhosis) at visit 1
7. renal dysfunction defined as glomerular filtration rate (GFR) < 60 mL/min/1.73 m2 at Visit 1
8. hypothyroidism that is not treated or not stable for at least 6 months prior to study entry
9. poorly controlled hypertension defined as a mean systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 100 mmHg at Visit 1. In individuals with end-organ damage, mean systolic blood pressure > 140 mmHg and mean diastolic blood pressure > 90 mmHg at Visit 1
10. severe hypotension defined as systolic blood pressure =< 90 mm Hg or diastolic blood pressure =< 60 mm Hg AND symptomatic
11. active peptic ulcer
12. known intolerance or allergy to niacin (nicotinic acid), niacinamide (nicotinamide), or any of the tablet ingredients: 1-methylnicotinamide chloride, microcrystalline cellulose, povidone, silicified microcrystalline cellulose, crospovidone, anhydrous dibasic calcium phosphate, hydroxypropyl cellulose, magnesium stearate (vegetable origin), polyvinyl alcohol, titanium dioxide, talc, polyethylene glycol, methacrylic acid copolymer, and sodium bicarbonate.
13. any known history of coronary artery disease, cerebrovascular disease or peripheral arterial disease
14. Use after screening to the conclusion of the study of any of the following lipid modifying medications/supplements:

    1. Niacin (nicotinic acid) or niacinamide (nicotinamide)
    2. Fibrates/fibric acid derivatives like fenofibrate, gemfibrozil, clofibrate
    3. Bile acid sequestrants like cholestyramine, colesevelam, colestipol
    4. HMG-CoA reductase inhibitors (statins) including atorvastatin, cerivastatin, fluvastatin, lovastatin, pravastatin, simvastatin, rosuvastatin
    5. Ezetimibe
    6. Omega-3 fatty acids
    7. Supplements containing flaxseed, tryptophan, fish oil, or algal oil.
    8. Sterol/stanol products
    9. Red yeast rice supplements or soy isoflavone supplements.
    10. Dietary fiber supplements including > 2 teaspoonfuls of Metamucil® or psyllium containing supplements per day.
    11. Other natural health products or prescription agents judged by the investigator to have the potential to alter serum lipid levels in an individual subject.
15. history of angina or myocardial infarction
16. hyperuricemia or with a history of gouty arthritis
17. known nephritic syndrome or >3 g protein/day in urine at Visit 1
18. known familial lipoprotein lipase deficiency, apo CII deficiency, or familial dysbetalipoproteinemia.
19. requirement for peritoneal dialysis or hemodialysis for renal insufficiency.
20. history of malignancy, except patients who have been disease-free for > 5 yrs, or resected basal or squamous cell skin carcinoma or cervical carcinoma in situ.
21. history of bariatric surgery.
22. history of pancreatitis, except secondary to cholelithiasis.
23. anticipation of major surgery during the study.
24. treatment with weight loss drugs or programs during the trial.
25. treatment with HIV-protease inhibitors, cyclophosphamide or isotretinoin.
26. treatment with tamoxifen, estrogens, or progestins that have not been stable for > 4 week prior to screening at Visit 1
27. routine or anticipated use of all systemic corticosteroids at Visit 1. Local, topical, inhaled, or nasal corticosteroids are permitted
28. blood donation of > pint (0.5 L) within 30 days prior to screening, or plasma donation within 7 days prior to screening at Visit 1
29. consumption of > 14 alcoholic drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor) at Visit 1.
30. history of drug abuse at Visit 1
31. participation in another clinical trial within 30 days of signing the information and consent form.
32. non-compliant to single blind investigational product (< 80% investigational product) or diet as per local judgment between Visit 1 and 4.
33. Any condition or therapy that the investigator believes might pose a risk or make participation in the study not in the patient's best interest.
34. Poor mental function or any reason to expect difficulty complying with the requirements of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  The number of patients randomized per site per month during the study
Compliance to investigational product | 14 weeks
  The proportion of randomized patients receiving the investigational product as per protocol.
Completion rate | 12 months
  The proportion of randomized patients completing the 14-week follow-up.

SECONDARY OUTCOMES:
Effect on serum high-density lipoprotein cholesterol (HDL-C) | 14 weeks
  The difference between groups in change from baseline to end of study in serum HDL-C.
Variability of serum triglycerides | 14 weeks
  The standard deviation of the change from baseline to end of study in serum triglycerides.
Effect on fasting glucose | 14 weeks
  The difference between groups in change from baseline to end of study in fasting glucose.
Effect on C-reactive protein | 14 weeks
  The difference between groups in change from baseline to end of study in C-reactive protein.
Effect on interleukin-6 (IL-6) | 14 weeks
  The difference between groups in change from baseline to end of study in IL-6.
Effect on total cholesterol (TC) | 14 weeks
  The difference between groups in change from baseline to end of study in TC
Effect on low-density lipoprotein cholesterol (LDL-C) | 14 weeks
  The difference between groups in change from baseline to end of study in LDL-C
Effect on very low-density lipoprotein cholesterol (VLDL-C) | 14 weeks
  The difference between groups in change from baseline to end of study in (VLDL-C),
Effect on total apolipoprotein B (apoB) | 14 weeks
  The difference between groups in change from baseline to end of study in apoB
Effect on total apolipoprotein A1 (apoA1) | 14 weeks
  The difference between groups in change from baseline to end of study in apoA1
Effect on lipoprotein (a) [Lp(a)] | 14 weeks
  The difference between groups in change from baseline to end of study in Lp(a)
Effect on non-high density lipoprotein cholesterol (non-HDL-C) | 14 weeks
  The difference between groups in change from baseline to end of study in non-HDL-C
Effect on TG/HDL-C ratio | 14 weeks
  The difference between groups in change from baseline to end of study in TG/HDL-C ratio
Effect on tumor necrosis factor - alpha (TNF-α) | 14 weeks
  The difference between groups in change from baseline to end of study in TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (17):
- Canada (17):
  - Crowfoot Village Family Practice, Calgary, Alberta
  - Dr. Senaratne Professional Corporation, Edmonton, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - Manna Research Vancouver, Vancouver, British Columbia
  - GA Research Associates, Ltd, Moncton, New Brunswick
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Scisco Clinical Research, Cornwall, Ontario
  - Sameh Fikry Medicine Professional Corp, Kitchener, Ontario
  - Aging, Rehabilitation & Geriatric Care, Lawson Health Research Institute-St Joseph's Health Care, Parkwood, London, Ontario
  - Prime Health Clinical Research, Toronto, Ontario
  - Manna Research Inc., Toronto, Ontario
  - Rhodin Recherche, Drummondville, Quebec
  - Recherche Invascor, Inc., Longueuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec, Inc., Québec, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Centre de santé et de services sociaux de Trois-Rivières, Trois-Rivières, Quebec